CLINICAL TRIAL: NCT03785847
Title: Normal Variability of Tidal Breathing Flow-volume Curves During Sleep in Healthy Children
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Revenio Research (Industry)
Responsible Party: Principal Investigator, Jussi Karjalainen, Head of Department, MD, PhD, Tampere University Hospital
Other Study IDs: VCS-008
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Respiration Disorders
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ventica — Impedance pneumography measurement

SUMMARY:
The study includes a comprehensive health examination with focus on respiratory health and the TBFV recordings using impedance pneumography (Ventica®) during sleep at night in healthy children.

DETAILED DESCRIPTION:
Impedance pneumograpy results in healthy children to generate normal values and to stude the effect of age and gender

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months-71 months, both sexes
* Healthy at the time of inclusion
* Signed informed consent

Exclusion Criteria:

* Preterm birth
* Recurrent bronchitis or recurrent hospitalizations because of a respiratory illness
* Nasal congestion, adenotonsillar hypertrophy, signs and symptoms of sleep apnea or sleep disordered breathing
* Acute respiratory infection or hospitalization because of an acute illness within 4 weeks prior to inclusion
* Personal or family history of asthma
* Recurrent wheezing without respiratory infection
* Allergic rhinitis, chronic rhinosinusitis, or other chronic respiratory disorders
* Atopic dermatitis
* Diagnosed allergic sensitization
* Use of asthma rescue or maintenance medication within 4 weeks prior to inclusion
* Any major chronic illness as judged by the investigators
* Implanted or external active medical devices such as pacemakers

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sample of 40 healthy children aged 12 - 71 months.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Ventica measurement | overnight measurement
  level of overnight tidal breathing flow volume variation

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Karjalainen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- TAYS Allergiakeskus, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seppa VP, Hyttinen J, Viik J. A method for suppressing cardiogenic oscillations in impedance pneumography. Physiol Meas. 2011 Mar;32(3):337-45. doi: 10.1088/0967-3334/32/3/005. Epub 2011 Feb 14. PMID 21321385
- [Background] Seppa VP, Hyttinen J, Uitto M, Chrapek W, Viik J. Novel electrode configuration for highly linear impedance pneumography. Biomed Tech (Berl). 2013 Feb;58(1):35-8. doi: 10.1515/bmt-2012-0068. PMID 23348215
- [Background] Seppa VP, Pelkonen AS, Kotaniemi-Syrjanen A, Makela MJ, Viik J, Malmberg LP. Tidal breathing flow measurement in awake young children by using impedance pneumography. J Appl Physiol (1985). 2013 Dec;115(11):1725-31. doi: 10.1152/japplphysiol.00657.2013. Epub 2013 Oct 3. PMID 24092693
- [Background] Malmberg LP, Seppa VP, Kotaniemi-Syrjanen A, Malmstrom K, Kajosaari M, Pelkonen AS, Viik J, Makela MJ. Measurement of tidal breathing flows in infants using impedance pneumography. Eur Respir J. 2017 Feb 15;49(2):1600926. doi: 10.1183/13993003.00926-2016. Print 2017 Feb. PMID 28182566
- [Background] Seppa VP, Pelkonen AS, Kotaniemi-Syrjanen A, Viik J, Makela MJ, Malmberg LP. Tidal flow variability measured by impedance pneumography relates to childhood asthma risk. Eur Respir J. 2016 Jun;47(6):1687-96. doi: 10.1183/13993003.00989-2015. Epub 2016 Mar 17. PMID 26989106